Timolol Eye Drops in the Treatment of Acute Migraine Headache NCT 02630719 4/22/19

## Statistical Analysis

The main outcome measure was percent of migraine attacks at 0 or 1 after treatment with timolol or artificial tears. A total of 198 migraine attacks were studied among 10 participants. The groups were compared using a Wilcoxon match paired test to account for repeated measurements and the difference between the two groups was found not to be significant. A 2-tailed chi-squared statistic suggested that 172 randomized participants would be needed to power a study with alpha </= 0.05 and beta </= 0.2.